CLINICAL TRIAL: NCT07322393
Title: Effect of Foot Reflexology On Chemotherapy Induced Nausea and Vomiting in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: Effect of Foot Reflexology On Chemotherapy Induced Nausea and Vomiting in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dania Azher Khan, MSN Student, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DAKhan
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an experimental group receiving foot reflexology in addition to standard care or a control group receiving standard care alone. Both groups will be followed in parallel throughout the study period.
Masking Description: This is an open-label study as blinding of participants and the researcher is not feasible due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Reflexology plus Standard Care (Experimental): Participants in this arm will receive foot reflexology in addition to standard chemotherapy care. Foot reflexology will be administered by the researcher using a standardized technique during chemotherapy sessions. Each session will last approximately 20-30 minutes and will be provided during each chemotherapy cycle with a 21-day interval. Standard care will be provided as per hospital protocol.
  Interventions: Other: Foot Reflexology
- Standard Care (No Intervention): Participants in this arm will receive standard chemotherapy care as per hospital protocol. No foot reflexology intervention will be provided.

INTERVENTIONS:
Other: Foot Reflexology — Foot reflexology is a complementary therapy involving the application of pressure to specific reflex points on the feet associated with nausea, vomiting, relaxation, and digestion. The intervention will be administered by the researcher for 20-30 minutes during chemotherapy sessions using a standardized technique.
  Arms: Foot Reflexology plus Standard Care

SUMMARY:
This study aims to evaluate the effect of foot reflexology on chemotherapy-induced nausea and vomiting in breast cancer patients. Nausea and vomiting are common side effects of chemotherapy and can negatively affect patients' comfort and quality of life. Foot reflexology is a non-invasive complementary therapy that involves applying pressure to specific points on the feet. The study will compare patients who receive foot reflexology along with standard care to those who receive standard care alone, to determine whether foot reflexology helps reduce the severity of nausea and vomiting during chemotherapy.

DETAILED DESCRIPTION:
This study will be conducted to assess the effectiveness of foot reflexology in reducing chemotherapy-induced nausea and vomiting among breast cancer patients receiving chemotherapy. Eligible participants will be adult breast cancer patients undergoing scheduled chemotherapy treatment.

After enrollment, participants will be randomly assigned into two groups: an experimental group and a control group. The experimental group will receive foot reflexology in addition to standard chemotherapy care, while the control group will receive standard care only.

Foot reflexology will be administered by the researcher using a standardized technique. Each session will last approximately 20-30 minutes and will be provided during chemotherapy sessions across multiple chemotherapy cycles with an interval of 21 days. Reflex points associated with nausea, vomiting, relaxation, and digestion will be stimulated using appropriate pressure techniques.

Nausea and vomiting will be assessed using a standardized assessment tool before and after the intervention during each chemotherapy cycle. The collected data will be analyzed to compare the severity of nausea and vomiting between the experimental and control groups to determine the effectiveness of foot reflexology as a supportive therapy for managing chemotherapy-induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer patients aged >18 Patients receiving chemotherapy in curative setting

Exclusion Criteria:

Patients with paraplegia. Patients with skin ulcers or wounds. Patients with psychiatric conditions. Patients with foot fractures and varicose veins. Patients with GIT and Liver Cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of Chemotherapy-Induced Nausea and Vomiting | From baseline to end of each chemotherapy cycle (up to four cycles, 21 days apart)
  The severity of chemotherapy-induced nausea and vomiting will be assessed using the Rhodes Index of Nausea, Vomiting and Retching (RINVR), a validated scale measuring the frequency, severity, and distress of nausea and vomiting. Scores range from low to high, with higher scores indicating more severe symptoms. Measurements will be recorded before and after the intervention during each chemotherapy cycle.

CONTACTS AND LOCATIONS:
Overall Officials: DR. Kausar Bano, MBBS, FCPS, Study Chair — Jinnah Hospital Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Article:Effect of Foot Reflexology on Chemotherapy Induced Nausea and Vomiting among Cancer Patients — https://journals.ekb.eg/article_293709_2ae2feb1a5ac3b48491377622893f2e3.pdf
- See also: Article:The Effect of Foot Reflexology on Chemotherapy Induced Nausea, Vomiting and Fatigue among Breast Cancer Patient — https://d1wqtxts1xzle7.cloudfront.net/107160937/The_20Effect_20of_20Foot_20Reflexology-libre.pdf?1699185869=&response-content-disposition=inline%3B+filename%3DThe_Effect_of_Foot_Reflexology_on_Chemot.pdf&Expires=1766409352&Signature=GuwXPqjLdyASok51kE1lzdUWTVRdOitwIpMdgl~xoaujhhxQuxY2yFH5wTQAFsVOUkT7NzJolPdBwgmqHPrxWbWCZG6z4yedV8yRX~vF9Vu3mFhIWGe3kPzkMQYuvM92LSvfwZZIHkVNk5q58z4WMbU34Ej3ysshDA-2xDboBenerJNKjVXnLVHvwWEt0zQvUwZ-h~bGdt2gHdOQIPceVzpEGn2d59cRwgWNE-jgiX3t4YLf~iyPvvduWxbk2xnHIqYZ1YGQzmU9UnfVL9~17AZSn7OvLp2MxvwbxYqTY5M7sXFQyY5ZyMc55nOkdxZHXWzuzQukA6UxC2XUstsv0g__&Key-Pair-Id=APKAJLOHF5GGSLRBV4ZA
- See also: Article: The Impact of Foot Reflexology on Nausea-Vomiting and Sleep Quality for Lung Cancer Patients Receiving Chemotherapy in Turkey — https://cyprusjmedsci.com/articles/the-impact-of-foot-reflexology-on-nausea-vomiting-and-sleep-quality-for-lung-cancer-patients-receiving-chemotherapy-in-turkey/doi/cjms.2022.2021-227